CLINICAL TRIAL: NCT05359471
Title: Characterization of Visceral Adiposity in HIV Mono-infected Patients With NAFLD
Acronym: Theratech
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Giada Sebastiani, Clinical Scientist at the Research Institute of McGill University, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-6656
Record Dates: First submitted 2022-04-22; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Visceral Steatosis; Hiv; NAFLD
MeSH Terms: conditions — Fatty Liver; Acquired Immunodeficiency Syndrome; Non-alcoholic Fatty Liver Disease | interventions — Absorptiometry, Photon; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: This is single center, cross sectional study conducted at the Chronic Viral Illness Service (CVIS) of McGill University Health Center (MUHC). This is a pilot feasibility study with the aim of further exploring more options to conduct or facilitate similar studies in larger group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV with NAFLD (Active Comparator): HIV Nonalcoholic fatty liver disease patients
  Interventions: Device: Bone densitometry; Other: Questionnaires; Device: Review of medical chart
- HIV without NAFLD (Active Comparator): HIV without Nonalcoholic fatty liver disease patients
  Interventions: Device: Bone densitometry; Other: Questionnaires; Device: Review of medical chart

INTERVENTIONS:
Device: Bone densitometry — It is the standard method for diagnosing osteoporosis. In the central DXA examination, which measures bone density of the hip and spine, the patient lies on a padded table.
  Other Names: Dual-energy x ray absorptiometry; DEXA; DXA
Other: Questionnaires — Smoking and drug related questionnaires will be used as variable to see dependence, how it impacts participants activities/health or determining whether they are light/moderate/heavy smoker
Device: Review of medical chart — History of previous liver diseases including hepatitis B, C, and HIV

SUMMARY:
To determine the distribution of visceral fat in people living with HIV (PLHIV) with NAFLD by clinical anthropometric indicators (wais-to-hip ratio), lipid accumulation product (waist circumference and triglycerides) and radiological techniques such as dual-energy X-ray absorptiometry (DXA) (trunk fat mass and fat mass through dual-energy X-ray absorptiometry).

DETAILED DESCRIPTION:
This is single center, cross sectional study conducted at the Chronic Viral Illness Service (CVIS) of McGill University Health Center (MUHC). This is a pilot feasibility study with the aim of further exploring more options to conduct or facilitate similar studies in larger group.. The investigator will correlate visceral fat with simple clinical parameters, including BMI and waist circumference and comparing measures of visceral fat between PLHIV with and without NAFLD. Participants will undergo a single study visit for confirmation of eligibility.

Until now, there has been no study assessing the distribution of visceral fat in PLHIV with NAFLD by clinical anthropometric indicators (WHR), lipid accumulation product (waist circumference, hip circumference and waist to hip ratio and triglycerides) and radiological techniques such as DXA. In the present feasibility pilot study, the investigator will determine the distribution of excessive fat around the abdomen(visceral fat) by DXA scan in HIV mono-infected patients with/without NAFLD to see if it will be possible to conduct a larger study.. The investigator will also correlate visceral fat with simple clinical parameters, including BMI and waist circumference and comparing measures of visceral fat between PLHIV with and without NAFLD.

DXA scan Bone densitometry, also called dual-energy x-ray absorptiometry, DEXA or DXA, uses a very small dose of ionizing radiation to produce pictures of the inside of the body (usually the lower (or lumbar) spine and hips) to measure bone loss. It is commonly used to diagnose osteoporosis, to assess an individual's risk for developing osteoporotic fractures. DXA is simple, quick and noninvasive. It's also the most commonly used and the most standard method for diagnosing osteoporosis.

Primary Objective

In order to determine if the distribution of visceral fat in PLHIV with NAFLD by clinical anthropometric indicators (waist-to-hip ratio), lipid accumulation product (waist circumference and triglycerides) and radiological techniques such as DXA (trunk fat mass and fat mass through dual-energy X-ray absorptiometry) could be used in future larger study groups.

Secondary Objectives

1. To correlate visceral fat with simple clinical parameters, including BMI and waist circumference.
2. To compare measures of visceral fat between PLHIV with and without NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old at screening;
* Able to provide informed consent, in French or English;
* Historical HIV seropositive (ELISA with Western blot confirmation);

Exclusion Criteria

* Contraindications to Fibroscan with CAP (pregnant women or individuals carrying a pacemaker);
* Historical evidence of co-infection with Hepatitis B or C (i.e. HBsAg or anti-HCV positive);
* Significant alcohol intake (>21 units/week in men and >14 units/week in women[23]) at screening using the Alcohol Use Disorders Identification Test (AUDIT-C) questionnaire;
* Patients with previous decompensating events from liver cirrhosis (Child-Pugh B and C), hepatocellular carcinoma, liver transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Determination of visceral fat | Through study completion, an average of 1 year
  Outcome Measures The primary outcome is the presence of high visceral fat, defined as >35% total body fat for females and >25% total body fat for males.

CONTACTS AND LOCATIONS:
Overall Officials: Giada Sebastiani, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada